CLINICAL TRIAL: NCT06181396
Title: Association Between Time of Oxytocin Initiation at 2nd Stage of Labor and Adverse Outcomes
Brief Title: Time of Oxytocin Initiation at 2nd Stage of Labor and Adverse Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Gal Bachar MD, Doctor of OBGYN, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0061-22-RMB
Record Dates: First submitted 2023-09-10; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Delivery Complication; Cesarean Delivery Affecting Fetus
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial of singleton gestations receiving oxytocin during the second stage of labor at a single tertiary medical center. Women will be randomly allocated to one of two groups - immediate initiation of oxytocin at full dilation versus delayed oxytocin initiation following one hour of full dilation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate oxytocin (Experimental): This arm will receive oxytocin when entering 2nd stage (full dilation)
  Interventions: Drug: Oxytocin
- Delayed oxytocin (Other): This arm will receive oxytocin one hour after entering 2nd stage (full dilation)
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Native oxytocin analog
  Other Names: Pitocin

SUMMARY:
Early oxytocin administration at the 2nd stage of labor is associated with a higher rate of vaginal delivery, shorter second stage duration, and fewer adverse maternal and neonatal outcomes.

DETAILED DESCRIPTION:
Cesarean delivery (CD) is one of the most common surgeries performed worldwide. In the last few decades, its rate has steadily increased worldwide, leading to an increase in maternal morbidity and mortality compared to vaginal delivery (VD)1. In 2014, the American College of Obstetricians and Gynecologists (ACOG) and Society for Maternal Fetal Medicine (SMFM) published an Obstetric Care Consensus for safe prevention of primary cesarean delivery, allowing an additional hour of pushing during the 2nd stage of labor for both nulliparous and multiparous women before diagnosing prolonged 2nd of labor2-4.

Prolonged 2nd stage is especially common among nulliparous women5, and is defined as more than three hours of pushing6, or four hours for women with a regional anesthesia. Prolonged 2nd stage has been shown to be associated with maternal adverse outcomes, such as assisted-vaginal delivery, CD, and postpartum hemorrhage (PPH)7,8, and neonatal adverse outcomes such as low 5-minute Apgar score, and NICU admissions9.

Oxytocin is the primary and the most widely used pharmacological agent for induction and augmentation of labor10. Administrating oxytocin during labor is a common practice and is used to intensify contractions and decrease the chances of a non-progressive labor and associated adverse outcomes11,12. Despite its extensive use, there are several protocols which varies between different countries and obstetric wards. Likewise, there is no consensus regarding the duration or dosage of oxytocin infusion during labor, and especially during the 2nd stage of labor13.

The study will assess the optimal time initiation of Oxytocin during the 2nd stage of labor, and its association to mode of delivery, and adverse maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy
2. Maternal age ≥ 18 years' old
3. Oxytocin administration initiated or renewed during second stage of labor

Exclusion Criteria:

1. Maternal age < 18 years' old
2. Multiple gestation pregnancy
3. Known fetal malformations
4. Uterine scar

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant Women
Enrollment: 120 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Mode of delivery | Delivery
  Vaginal or instrumental or cesarean

SECONDARY OUTCOMES:
2nd stage duration | Delivery
  Minutes
intrapartum fever | Delivery or 48 hours postpartum
  Rate of chorioamnionitis
Meconium stain | Delivery
  Rate
Postpartum hemorrhage | Delivery
  more than 500 ml following vaginal delivery or more than 1000 ml at cesarean delivery
FHR decelerations | Delivery
  Variable or Late Decelerations viewed by the physician according to external fetal monitor.
Neonatal pH | Delivery
  Umbilical cord pH
Neonatal Apgar score | Delivery
  5 minutues Apgar score
Admission of the neonate to neonatal intensive care unit | Immediate postpartum, up to 5 days.
  Admission of the neonate to neonatal intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam medical health campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes